CLINICAL TRIAL: NCT04648813
Title: Tiotropium Efficacy Against Allergen Induced Early Asthmatic Responses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Beth Davis, Research Scientist, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO REB 1959
Record Dates: First submitted 2020-11-23; First posted 2020-12-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Allergic Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tiotropium bromide monohydrate (Spiriva Respimat) (Experimental)
  Interventions: Drug: tiotropium bromide monohydrate (Spiriva Respimat)
- matching placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: tiotropium bromide monohydrate (Spiriva Respimat) — administered daily, 2 inhalations/5mcg per dose for a total of 8 doses
  Arms: tiotropium bromide monohydrate (Spiriva Respimat)
Drug: matching placebo — administered daily, 2 inhalations per dose for a total of 8 doses
  Arms: matching placebo

SUMMARY:
The study will compare the effect of inhaled tiotropium versus placebo on allergen induced early asthmatic responses in individuals with atopic asthma.

DETAILED DESCRIPTION:
This is a single center, double-blind, randomized, placebo-controlled, crossover study. The study will consist of two one week treatment periods, one with tiotropium (two inhalations/5mcg/day) and one with placebo (2inhalations/day). A minimum two week washout period between treatments is required. Four visits over the course of approximately 4 weeks will be required to complete the study. Procedures at each visit are as follows:

Visit 1:

Participants will undergo consent procedures and if consent is provided measurements of FeNO, spirometry, airway responsiveness to methacholine, skin prick testing, skin titration endpoint testing and sputum induction will be performed. If participants meet eligibility criteria following these assessments, treatment 1 will be dispensed and the first dose administered. The participant will then self administer the treatment for the next six days (i.e. a total of 7 days of treatment) before returning for Visit 2.

Visit 2:

A final dose of treatment 1 will be administered. At 30 minutes post dose, FeNO testing, spirometry measurements and allergen inhalation challenge will be performed. Five hours after the allergen challenge, FeNO will again be measured and sputum induction will be performed.

Visits 3 and 4:

Visits 3 and 4 will be identical to Visit 1 and 2 except that no skin prick testing or skin titration endpoint testing will be required. At Visit 3 participants will be crossed over to treatment 2 and the first dose will be administered. Participants will self administer treatment 2 for the next six days before returning for Visit 4.

The primary endpoint will be the EAR PD20, the amount of allergen required to induce an early asthmatic response (i.e. a fall in FEV1 post allergen inhalation of 20% or more) tiotropium versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosis of mild asthma with a minimum 3 months history at the time of enrolment into the trial
* pre-bronchodilator FEV1 80% or greater than the predicted value
* positive response to inhaled methacholine (i.e. MCh PD20 ≤ 400mcg)
* evidence of atopy (i.e. positive skin prick test to an allergen that is appropriate for use in allergen inhalation challenge)
* no respiratory infection within 4 weeks of Visit 1
* no allergen exposure within 4 weeks of Visit 1
* current non-smoker (ex-nicotine smoker with < 10 pack years evaluated case by case)
* use of β2 agonist rescue medications less than daily and no more than 4 times per week
* general good health with no other medical condition, medication use or lifestyle activities that would potentially alter the outcome of the allergen challenge

Exclusion Criteria:

* currently pregnant or breast-feeding
* current daily use of other inhaled recreational products (e.g. cannabis, e-cigarettes or other vaping products; occasional use requires 24 hour withhold)
* diagnosis or evidence of narrow angle glaucoma
* diagnosis or evidence of urinary retention
* known hypersensitivity to tiotropium, atropine or its derivatives (e.g. ipratropium) or components of tiotropium formulation (e.g. benzalkonium chloride)
* history of anaphylaxis or angioedema
* current use of :
* inhaled corticosteroid including combination therapies
* inhaled muscarinic antagonists - except study treatment (e.g. ipratropium bromide)
* long-acting beta2-agonists (LABA; e.g. formoterol)
* leukotriene receptor antagonists (e.g. montelukast)
* biologics (e.g. benralizumab)
* allergen immunotherapy
* mast cell stabilizers (e.g. nedocromil sodium)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
EAR PD20 | 30 minutes post last dose of treatment
  amount of inhaled allergen required to induce a 20% fall in FEV1

SECONDARY OUTCOMES:
Airway inflammation | pre-treatment, 30 minutes post final dose and 5 hours post allergen inhalation challenge
  level of FeNO (fractional exhaled nitric oxide) in parts per billion (ppb)
Airway inflammation | pre treatment and 5 hours post allergen inhalation challenge
  change in number of sputum differential cell counts, specifically eosinophils

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma Research Lab University of Saskatchewan Room 346 Ellis Hall, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No